CLINICAL TRIAL: NCT01025362
Title: Baby-Friendly Community Health Services Evaluation: A Cluster Randomised Controlled Study
Brief Title: Baby-Friendly Community Health Services Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Berug, director, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S-09277c2009/5783
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactation counseling (Experimental): Intervention arm: The mother and child health centres will implement The Baby-Friendly Initiative to improve their lactation counseling.
  Other Names: The Baby Friendly Community Health Service
  Interventions: Behavioral: Lactation counseling
- Standard care (Active Comparator): The comparison group was mother and child health centres which continued offering standard care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Lactation counseling — The Baby-Friendly Community Health Service intervention to improve quality of lactation counseling.
  Other Names: The Baby-Friendly Community Health Service
  Arms: Lactation counseling
Behavioral: Standard care — Child Health Services offered standard care
  Arms: Standard care

SUMMARY:
The Norwegian Action Plan on Nutrition aim at increasing the prevalence of breastfeeding. The initiative "Baby-Friendly Community Health Services (BFCHS)" is an initiative to reach this goal. BFCHS is developed from the concept "The Baby-Friendly Hospital Initiative" by WHO/UNICEF, and the intention is to increase the quality of breastfeeding counseling at Norwegian well-baby clinics.

The purpose of the study

The study seeks to answer the following research questions:

* What effect does the process of being certified as a BFCHS have on the proportion of mothers who exclusively breastfeed their children for 5 months?
* What effect does the process of being certified as a BFCHS have on the proportion of mothers who exclusively breastfeed for 4 months?
* What effect does the certification process have on the proportion of mothers who breastfeed at 11 months of age?
* What effect does the certification process have on the differences in breastfeeding due to social inequality?
* What effect does the certification process have on the mothers impression of the quality of the well-baby clinics lactation counseling?
* What effect does the certification process have on mothers satisfaction with the breastfeeding experience?
* What effect does the certification process have on perceived pressure to breastfeed? Methods Cluster randomized controlled study Sampling The survey unit, cluster, will be the community health services. All community health services in six counties in Norway will be invited to participate.

Inclusion criteria: Norwegian speaking mothers who have 5 month and 11 month old children.

Data collection Respondents are identified through the National Population Register (DSF). The data collection takes place using a postal questionnaire.

Baseline: Data collection before the intervention is implemented to assess breastfeeding prevalence and distribution of covariates in the two study arms.

Post-survey: The post-survey to assess the effect, will take place about two years after baseline when the community health services have been certified.

Sample size It is expected that the project could increase the breastfeeding prevalence with 5 percentage points. This assumption is the basis for the sample size. The initial aim is to recruit about 50 well-baby clinics.

DETAILED DESCRIPTION:
In 2007 the Norwegian Government launched "The Norwegian Action Plan on Nutrition" (2007-2011) which emphasizes breast milk as optimal nutrition as well as being one of the most effective ways to promote health and prevent disease. It is well known that breast milk reduces the prevalence and severity of infectious diseases like diarrhoea, lower respiratory tract infections, ear infections, urinary tract infections as well as bacterial meningitis and necrotic enterocolitis. Current research suggests that breast milk can have long term health effects such as reduced risk of overweight, leukemia and diabetes type I and type II. Breastfeeding is associated with better cognitive development. Women who breastfeed also have significant added health benefits such as a reduced risk of breast cancer.

Almost all women produce breast milk, but the act of breastfeeding is a complicated interaction between mother and child and is affected by a number of factors. A large number of mothers have breastfeeding difficulties, and a significant number stop before they had intended to. If women were given qualified help it is possible that many of these problems could have been prevented or treated. In the Norwegian subsidiary study to The WHO Multicentre Growth Reference Study, where mothers received qualified breastfeeding instruction, 86% of children were exclusively breastfed at the 4 month stage as compared with the norm of 44%.

Today mothers are discharged earlier from hospital than ever before. Many of these women have not managed to properly establish breastfeeding. Due to this, many problems which were previously discovered in the maternity ward are now relegated to the primary health care services.

The disparity in breastfeeding between different socioeconomic groups in Norway primarily follows the same pattern as that found in health generally.For example, the chance that a mother with higher education will be breastfeeding her child at the age of 6 months is twice as high compared to a mother with only primary school education. Improving health service access to the entire population would contribute to advancing the health and health promoting behavior in those groups with the poorest prospects.

The National Resource Centre for Breastfeeding (NRCB) is cooperating with Norwegian Public Health Nurses Association and the Norwegian Directorate of Health in the initiative Baby-Friendly Community Health Services (BFCHS). The purpose of this initiative is to improve the quality of breastfeeding advice at Norwegian community health services.

While WHO has developed an international standard for breastfeeding counseling for maternity wards, there is no similar standard for primary care services as yet.

A newly updated Cochrane-overview about the effect of offering support to breastfeeding mothers identified 16 studies which assessed the effect of support from health workers. The studies showed a small effect on all breastfeeding at the four month stage, but could not show any difference at other stages. An American survey identified 38 randomized controlled studies on the effect of initiatives in primary care services to promote breastfeeding, all from industrialized countries.This review indicates that initiatives to increase the competency of health workers can have a positive effect on the prevalence of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with infants of five and eleven months age.
* Mothers who are able to understand Norwegian.

Exclusion Criteria:

* Mothers who do not understand Norwegian.
* Mothers with infants below five months and above twelve months age.

Ages: 5 Months to 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2032 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding prevalence | infants age: five months

SECONDARY OUTCOMES:
Exclusive breastfeeding prevalence | infants age: 4 months
Any breastfeeding prevalence | infants age: 5 months and 11 months
Mothers perception of quality of lactation counselling | infants age: 5 months
Mothers satisfaction with the breastfeeding experience | Infants age: 6 months
Mothers perception of breastfeeding pressure | Infants age: 6 mon

CONTACTS AND LOCATIONS:
Overall Officials: Beate F Loland, Md PhD, Principal Investigator
Locations (1):
- Rikshospitalet HF, Oslo, Norway

REFERENCES:
- [Derived] Baerug A, Laake P, Loland BF, Tylleskar T, Tufte E, Fretheim A. Explaining socioeconomic inequalities in exclusive breast feeding in Norway. Arch Dis Child. 2017 Aug;102(8):708-714. doi: 10.1136/archdischild-2016-312038. Epub 2017 Feb 24. PMID 28235835